CLINICAL TRIAL: NCT05079009
Title: Effects of Blood Pulsatility on Von Willebrand Factor During Extracorporeal CO2 Removal (ECCO2R)
Brief Title: Effects of Blood Pulsatility on Von Willebrand Factor During ECCO2R
Acronym: FLOW-ECCO2R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Xenios AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP180481; DR-2020-302 (Other: Commission Nationale de l'Informatique et des Libertés); 2020-A00156-33 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2021-07-31; First posted 2021-10-15 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Extracorporeal CO2 Removal; Acute Respiratory Distress Syndrome; Chronic Obstructive Pulmonary Disease Exacerbation; Pulmonary Disease
Keywords: ECCO2R; Willebrand factor; ARDS; COPD
MeSH Terms: conditions — Respiratory Distress Syndrome; Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECCO2R pulsatile configuration (Experimental): Adult patients hospitalized in the medical ICU for whom a treatment by ECCO2R has been indicated.
  Interventions: Device: ECCO2R pulsatile configuration

INTERVENTIONS:
Device: ECCO2R pulsatile configuration — Use of the pulsatile extracorporeal blood flow configuration.

SUMMARY:
The primary objective of the study is to demonstrate that the ECCO2R pulsatile configuration prevents the Willebrand factor high molecular weight multimers decrease observed under continuous blood flow configurations.

The secondary objectives are to quantify the CO2 extracorporeal removal in the pulsatile configuration, to describe complications (hemorrhagic, thrombotic and hemolytic), to describe patients' gas exchanges under ECCO2R, to describe the clinical course of the patients under ECCO2R as well as during the whole stay in the Intensive Care Unit (ICU).

DETAILED DESCRIPTION:
A track of major interest to prevent bleeding complications in ECCO2R, and more generally in extracorporeal circulations, is to prevent acquired Willebrand disease. Indeed, a loss of Willebrand factor high molecular weight multimers (Whmwm) is frequently observed in conditions characterized by a continuous blood flow, associated with a high incidence of bleeding. A publication suggested the existence of this phenomenon under ECCO2R achieved through the medical device Hemolung (Alung technology, USA). We preliminary observed an almost constant and early (< 24 hours) decrease in Willebrand factor high molecular weight multimers under ECCO2R. Such a phenomenon is considered as a major factor of hemorrhagic complications. We hypothesize that use of pulsatile extracorporeal blood flow configuration during the full length of ECCO2R therapy, as authorized by the Xenios console (Xenios AG, Heilbronn), would preserve a normal value of Whmwm, mainly by changing the conditions of shear constraints ("shear stress").

ELIGIBILITY:
Inclusion Criteria:

* Adult patient hospitalized in the Georges Pompidou European Hospital medical ICU
* Patient with or without SARS-CoV-2 infection
* ECCO2R treatment decision made by the medical team (regardless of the FLOW-ECCO2R protocol): mainly ECCO2R to enable ultraprotective ventilation for Acute respiratory distress syndrome (ARDS) patients or to avoid intubation or to shorten invasive mechanical ventilation in Chronic obstructive pulmonary disease (COPD) patients
* Affiliation to a social security regimen
* Informed consent (patient, trusted person, close family) , by default emergency inclusion notified in medical file and pursuance consent sought
* Negative serum or urinary β-hCG for women of child-bearing potential

Exclusion Criteria:

* Known allergy to heparin or to any of the excipients of the specialty used
* History of type II heparin-induced thrombopenia
* Thrombocytopenia (platelet < 100.000/mm3)
* Constitutional hemostasis disease interfering with biological assays
* Organic lesion likely to bleed
* Bleeding manifestations or tendencies linked to disorders of hemostasis
* Intracerebral hemorrhage
* Participation in another interventional research involving human participants
* Pregnant or breastfeeding women
* Protected adults (including individual under guardianship by court order)
* Persons deprived of their liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Level course of Willebrand Factor high molecular weight multimers in plasma | Up to 30 days
  Quantification of plasma Willebrand Factor high molecular weight multimers by the Hydrasys system

SECONDARY OUTCOMES:
Rate of specific adverse events | Up to 30 days
  To describe the complications under ECCO2R: hemorrhagic, thrombotic and hemolytic adverse events
Level of von Willebrand factor | Up to 30 days
  To quantify von Willebrand activity/antigenemy
Level of P-Selectin | Up to 30 days
  Characterization of the blood coagulation system
Level of leucoplatelet aggregates | Up to 30 days
  Characterization of the blood coagulation system
Level of proplatelet aggregates | Up to 30 days
  Characterization of the blood coagulation system
Level of platelet | Up to 30 days
  Characterization of the blood coagulation system
Level of microparticles | Up to 30 days
  Characterization of the blood coagulation system
Level of leucocytes | Up to 30 days
  Characterization of the blood coagulation system
Level of endothelial cells | Up to 30 days
  Characterization of the blood coagulation system
Level of NETs (Neutrophil Extracellular Traps) | Up to 30 days
  Characterization of the blood coagulation system
Level of free DNA | Up to 30 days
  Characterization of the blood coagulation system
Level of Nucleosome | Up to 30 days
  Characterization of the blood coagulation system
Level of FiO2 | Up to 29 days
  Recording of mechanical ventilator parameters (Non-Invasive Ventilation or Invasive Mechanical Ventilation) to describe the patients' clinical course under ECCO2R as well as during the whole stay in the ICU.v
VT (Tidal Volume) | Up to 29 days
  Recording of mechanical ventilator parameters (Non-Invasive Ventilation or Invasive Mechanical Ventilation) to describe the patients' clinical course under ECCO2R as well as during the whole stay in the ICU.v
Respiratory rate | Up to 29 days
  Recording of mechanical ventilator parameters (Non-Invasive Ventilation or Invasive Mechanical Ventilation) to describe the patients' clinical course under ECCO2R as well as during the whole stay in the ICU.v
Level of PaO2 | Up to 29 days
  Description of the arterial blood gas parameters under ECCO2R
Level of PaCO2 | Up to 29 days
  Description of the arterial blood gas parameters under ECCO2R
pH | Up to 29 days
  Description of the arterial blood gas parameters under ECCO2R
Level of SaO2 | Up to 29 days
  Description of the arterial blood gas parameters under ECCO2R
Heart rate | Up to 30 days
  To describe the patient vital parameters under ECCO2R
Respiratory rate | Up to 30 days
  To describe the patient vital parameters under ECCO2R
Blood Pressure | Up to 30 days
  To describe the patient vital parameters under ECCO2R
Pump speed | Up to 29 days
  Description of the ECCO2R parameters
Pulsatility setting | Up to 29 days
  Description of the ECCO2R parameters
Extracorporal blood flow | Up to 29 days
  Description of the ECCO2R parameters
Extracorporal pressures | Up to 29 days
  Description of the ECCO2R parameters

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Diehl, PhD, Study Chair — AP-HP, Hôpital Européen Georges Pompidou, Paris
Locations (1):
- Hôpital européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Kalbhenn J, Neuffer N, Zieger B, Schmutz A. Is Extracorporeal CO2 Removal Really "Safe" and "Less" Invasive? Observation of Blood Injury and Coagulation Impairment during ECCO2R. ASAIO J. 2017 Sep/Oct;63(5):666-671. doi: 10.1097/MAT.0000000000000544. PMID 28187047